CLINICAL TRIAL: NCT04562259
Title: Verification of Kimmerle's Anomaly by X-ray Methods of Research
Status: Active, not recruiting | Type: Observational
Sponsor: Samarkand State Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Project#3
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Kimmerle's Anomaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Kimmerle's anomaly: patients who have a complete or incomplete bony bridge over the posterior arch of the first cervical vertebra
  Interventions: Radiation: Verification of Kimmerle's anomaly by x-ray methods of research

INTERVENTIONS:
Radiation: Verification of Kimmerle's anomaly by x-ray methods of research — In patients with Kimmerle's anomaly, using computed tomography of the brain with the capture of the upper cervical spine and cervical spine, it is planned to determine at what age this pathology is more common, localization of the anomaly (right, left), complete or incomplete form of the anomaly.

SUMMARY:
Kimmerle's anomaly is a bony bridge over the posterior arch of the first cervical vertebra that forms a bony ring. The vertebral artery passes through the opening. This bone bridge could theoretically be an extravasal compression of the artery and disrupt the normal blood flow to the brain. Evaluating the data of X-ray methods, determine the frequency of occurrence and types of Kimmerle anomaly.

DETAILED DESCRIPTION:
It is planned to conduct an examination of 30 patients on the basis of the Department of Radiation Diagnostics and Therapy of the Samarkand State Medical Institute. Patients of all ages will be examined, directed by doctors for computed tomography of the brain with the capture of the upper cervical spine and the cervical spine. with complaints of headache, dizziness, pain in the cervical region Among those who have passed the study, it is necessary to identify patients with Kimmerle's anomaly and determine the age at which it often occurs, whether it is a congenital pathology or the result of degenerative-dystrophic changes. It is also planned to calculate the frequency of occurrence among the population, the type of this pathology (complete and incomplete bone bridge, right-sided and left-sided location), the size of the hole formed. The condition of the posterior parts of the brain will be assessed in the presence of Kimmerle's anomaly on a CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Kimmerle's anomaly

Exclusion Criteria:

* patients in whom the structure of the first cervical vertebra is not clearly visible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages will be examined, directed by doctors for computed tomography of the brain with the capture of the upper cervical spine and the cervical spine. with complaints of headache, dizziness, pain in the cervical region
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
In patients with Kimmerle anomaly, determine the types of forms of this pathology | up to 36 months
  In patients with Kimmerle's anomaly, using computed tomography of the brain with the capture of the upper cervical spine and cervical spine, it is planned to determine at what age this pathology is more common, localization of the anomaly (right, left), complete or incomplete form of the anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Gulshod Mardieva, docent, Study Director — Samarkand State Medical Institute
Locations (1):
- Samarkand State Medical Institute, Samarkand, Uzbekistan